CLINICAL TRIAL: NCT01004510
Title: An Open-Label Phase II Study of Zometa as Adjuvant Treatment of Malignant Pleural Effusion Due to Non-Small Cell Lung Cancer
Brief Title: Zometa Adjuvant Treatment of Malignant Pleural Effusion Due To Non-Small Cell Lung Cancer
Acronym: ZAP
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: failure to accrue projected number of patients
Sponsor: Peter Bushunow MD (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Peter Bushunow MD, Director, Oncology Research, Rochester General Hospital
Organization: Rochester General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: US CZOL446EUS143T
Record Dates: First submitted 2009-10-29; First posted 2009-10-30 (Estimated); Results first posted 2012-12-04 (Estimated); Last update posted 2012-12-04 (Estimated); Status verified 2012-11

CONDITIONS: Malignant Pleural Effusion; Non Small Cell Lung Cancer
Keywords: malignant pleural effusion; non small cell lung cancer
MeSH Terms: conditions — Pleural Effusion, Malignant; Carcinoma, Non-Small-Cell Lung | interventions — Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Zoledronic Acid (Experimental): Zometa administered as a 15 minute IV infusion of either 4 mg, 3.5mg, 3.3 mg or 3.0 mg every 4 weeks based on the patient's baseline calculated creatinine clearance(CrCl)using the Cockcroft-Gault formula.
  Interventions: Drug: zoledronic acid

INTERVENTIONS:
Drug: zoledronic acid — Zoledronic acid (Zometa) 4mg IV every 4 weeks for 3 treatments with chemotherapy as selected by treating physician
  Other Names: Zometa

SUMMARY:
The purpose of this study is to evaluate whether the addition of the bisphosphonate Zometa (zoledronic acid) used along with standard regimens of chemotherapy, will help to control the need for palliative intervention of malignant pleural effusions due to non-small cell lung cancer.

DETAILED DESCRIPTION:
Malignant pleural effusions are common in late stage non-small cell lung cancer and can lead to significantly increased morbidity in this patient population. The majority of patients are symptomatic due to their malignant effusions. The recurrence rates are thought to be quite high overall and may approach 100% without any further treatment.Currently there is no available non-invasive, medical means for controlling the effusions other than systemic chemotherapy.Zoledronic acid has been shown in a mouse model of malignant pleural effusion to decrease fluid accumulation and tumor dissemination while prolonging survival.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented non-small cell lung cancer, Stages 3B, 4 or recurrent
* Pleural effusion cytologically proven to be malignant
* 0 or 1 prior chemotherapy regimens for non-small cell lung cancer (adjuvant chemotherapy post resection, or concurrent chemo-radiation therapy counts as one regimen regardless of number of agents used.)
* Planning to start chemotherapy for non-small cell lung cancer (treatment regimen at discretion of treating physician but must include one or more of the following agents:cisplatin,carboplatin,docetaxel,paclitaxel, pemetrexed,gemcitabine,vinorelbine) Patients may receive anti-angiogenesis agents (bevacizumab) in addition to chemotherapy, but patients treated solely with tyrosine kinase inhibitors or growth-factor receptor blockers are not eligible.
* Prior radiation therapy is permitted.
* Performance status 0,1,2
* Serum creatinine less than 2.0 or estimated creatinine clearance over 30cc/min by Calcroft/Gault equation
* Estimated life expectancy over 3 months
* Signed informed consent
* Age greater than 18 years
* Patients who have clinical indication for Zometa treatment such as lytic bone metastases or hypercalcemia can be included

Exclusion Criteria:

* Pregnant or lactating
* Patient with concurrent medical or psychiatric illness which would, in the opinion of the investigator, prevent compliance with the study
* Patients who undergo any procedure other than thoracentesis for drainage of effusion.Patients may have had more than one thoracentesis prior to study. Patients who have large bore chest tube placement, permanent transthoracic catheter (Pleurex), medical pleurodesis or thoracoscopy are excluded.
* Current active dental problems including infection of the teeth or jawbone (maxilla or mandibular);dental or fixture trauma, or a current or prior diagnosis of osteonecrosis of the jaw (ONJ), of exposed bone in the mouth, or of slow healing after dental procedures.
* Recent (within 6 weeks)or planned dental or jaw surgery (e.g.extraction, implants).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2009-11; Primary Completion 2010-09 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Todd Sheppard, M.D., Principal Investigator — Rochester General Hospital; Peter Bushunow, M.D., Principal Investigator — Rochester General Hospital; Kevin Lightner, M.D., Principal Investigator — Rochester General Hospital
Locations (1):
- Rochester General Hospital, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Zoledronic Acid: Monthly zoledronic acid in addition to chemotherapy. Zoledronic acid dose per package insert for up to 4 cycles.
Period: Overall Study
Arm/Group | Zoledronic Acid
Started | 3
Completed | 2
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Groups:
- Zoledronic Acid: Monthly zoledronic acid in addition to chemotherapy
Arm/Group | Zoledronic Acid
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 3
control of malignant pleural effusions in non small cell lung cancer [Number; unit: participants] | 3

OUTCOME MEASURES:

1. Primary Outcome: Rate of Control (Lack of Need for Palliative Intervention of Malignant Pleural Effusions) in Patients With Non Small Cell Lung Cancer Treated With Standard Regimens of Cytotoxic Chemotherapy With the Addition of Zometa
Time Frame: 3 months
Population: Too few patients enrolled to analyze data
Arm/Group | Zoledronic Acid
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Although the protocol was approved to begin enrollment 9/25/09, Adverse event data was collected from first patient enrollment 1/4/10-through study termination on 4/26/11. Aproximately 1 year, 4 months.
Arm/Group | Zoledronic Acid
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 1/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zoledronic Acid (N=3)
Admitted to hospital with diagnosis of pneumonia and anemia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zoledronic Acid (N=3)
erythematous prurtic rash over chest and abdomen (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes